CLINICAL TRIAL: NCT06412926
Title: A Crossover Treatment, Phase 1, Open-label, Relative Bioavailability Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Single Doses of 2 Formulations of Emodepside (BAY 44-4400), and to Assess the Effect of Food in Healthy Male and Female Participants.
Brief Title: A Study to Learn About How Much Emodepside Gets Absorbed in the Blood and How Food Affects Its Absorption When Given as a New Type of Tablet to Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 22534; 2023-508905-26-00 (Other: EMA - EU CT Number)
Record Dates: First submitted 2024-05-02; First posted 2024-05-14 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Soil-transmitted Helminth Infection; Onchocerciasis (River Blindness)
Keywords: Soil-transmitted helminth infection; Onchocerciasis (river blindness)
MeSH Terms: conditions — Onchocerciasis; Onchocerciasis, Ocular | interventions — Bay 44-4400

STUDY DESIGN:
Intervention Model Description: The study will be conducted in a single-center, randomized, open label, cross over design.
  The study will investigate the relative bioavailability, pharmacokinetics, safety and tolerability of single doses of 2 formulations of emodepside and assess the effect of food on Test formulation (Formulation B) in healthy male participants and healthy female participants of non-childbearing potential.
  The crossover design is used for intra-individual comparison of treatment effects to reduce impact of inter-individual variability. A preliminary PK analysis is planned after Period 2 to determine the appropriate dose to be tested for food effect.
  Treatment allocation is conducted in a randomized manner prior to Period 1 in order to reduce the likelihood of period or seasonal effects confounding the study assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Period 1 Formulation A, fasted (Experimental): All subjects will receive either Formulation A or Formulation B per randomisation scheme as a single dose in fasted state.
  Interventions: Drug: BAY 44-4400
- Period 1 Formulation B, fasted (Experimental): All subjects will receive either Formulation A or Formulation B per randomisation scheme as a single dose in fasted state.
  Interventions: Drug: BAY 44-4400
- Period 2 - Crossover Formulation A, fasted (Experimental): All subjects will receive either Formulation A or Formulation B Cross-over: dependent on what they received in period 1 per randomisation scheme as a single dose in fasted state
  Interventions: Drug: BAY 44-4400
- Period 2 - Crossover Formulation B fasted (Experimental): All subjects will receive either Formulation A or Formulation B Cross-over: dependent on what they received in period 1 per randomisation scheme as a single dose in fasted state
  Interventions: Drug: BAY 44-4400
- Period 3 - no dose adjustment after Period 2 (Experimental): If no dose adjustment was needed after Period 2, all subjects will receive Formulation B in fed state
  Interventions: Drug: BAY 44-4400
- Period 3 - dose adjustment after Period 2, fasted (Experimental): If dose adjustment was needed after period 2, all subjects will receive Formulation B as single dose either in fasted or in fed state
  Interventions: Drug: BAY 44-4400
- Period 3- dose adjustment after Period 2, fed (Experimental): If dose adjustment was needed after period 2, all subjects will receive Formulation B as single dose either in fasted or in fed state
  Interventions: Drug: BAY 44-4400
- Period 4 - crossover following Period 3 (in case of dose adjustment after Period 2), fasted (Experimental): All subjects will receive Formulation B as single dose either in fasted or in fed state depending on if they were in the fasted or fed group in Period 3
  Interventions: Drug: BAY 44-4400
- Period 4 - crossover following Period 3 (in case of dose adjustment after Period 2), fed (Experimental): All subjects will receive Formulation B as single dose either in fasted or in fed state depending on if they were in the fasted or fed group in Period 3
  Interventions: Drug: BAY 44-4400

INTERVENTIONS:
Drug: BAY 44-4400 — Film-coated tablet, oral use
  Other Names: Formulation A
  Arms: Period 1 Formulation A, fasted; Period 2 - Crossover Formulation A, fasted
Drug: BAY 44-4400 — Film-coated tablet, oral use
  Other Names: Formulation B
  Arms: Period 1 Formulation B, fasted; Period 2 - Crossover Formulation B fasted; Period 3 - dose adjustment after Period 2, fasted; Period 3 - no dose adjustment after Period 2; Period 3- dose adjustment after Period 2, fed; Period 4 - crossover following Period 3 (in case of dose adjustment after Period 2), fasted; Period 4 - crossover following Period 3 (in case of dose adjustment after Period 2), fed

SUMMARY:
Onchocerciasis or river blindness is an infectious disease caused by a parasitic worm. It spreads through the bite of an infected blackfly. Common symptoms include severe itching, skin problems, and eye problems including permanent blindness.

Soil-transmitted helminthiasis is an infection caused by various parasitic worms, such as whipworm, hookworm, and roundworm in the intestines. The infection spreads through eggs found in the feces of infected people. This contaminates the soil in areas with poor sanitation. Common symptoms include stomach pain, loose stools, loss of blood and proteins, delayed development in children, and reduced work performance in adults.

Researchers are looking for better ways to treat onchocerciasis and soil-transmitted helminthiasis. Emodepside is being tested for the treatment of onchocerciasis and soil-transmitted helminthiasis in both men and women. It works by activating a protein called 'SLO-1', which causes paralysis and death of the parasitic worms.

The main purpose of this study is to find out if there is a difference in how emodepside gets absorbed in the blood when given as a new tablet compared to the existing tablet, as a single dose. Researchers also want to find the effect of food on the absorption of the new emodepside tablet.

The amount of emodepside in participants' blood will be measured at various time points. These will be used to calculate and compare the following measurements after a single dose of the new and existing tablet of emodepside without food.

The amount of emodepside in participants' blood will be measured at various time points. These will be used to calculate the Cmax and AUC after a single dose of the new tablet of emodepside with and without food. The number of participants who experience medical problems during this study will be documented.

During this study, participants will receive 2 different types of emodepside tablets. These include the newly developed tablet and an existing tablet that has already been used in other clinical studies.

At the start of the study, the researchers will ask participants about their medical and surgical history. They will also perform a health check-up for all participants, and pregnancy tests for women.

During the study, participants will have blood and urine samples taken to check for any medical problems and to measure the amount of emodepside in the blood.

The study doctors will confirm that the participants can take part in the study. This may take up to 21 days.

This study has 3 or 4 periods and contains up to 2 in-house periods of 16 days each.

On Day 1 of each period, participants will receive the treatments, but the order of the treatment will be different.

• Periods 1 and 2: Each participant will receive a single oral dose of the new or the existing emodepside tablet without food.

After Period 2, an initial analysis will be performed. This analysis will help decide the doses for the next periods.

* Period 3: Participants will receive a selected dose of the new emodepside tablet either with or without food.
* Period 4 (optional): If needed, participants may receive a selected dose of the new emodepside tablet either with or without food. The decisions to conduct Period 4 will depend on the results of the initial analysis.

Participants will have a total of 6 additional weekly visits to the study site for sample collection after the last period (either Period 3 or 4).

Participants will attend a follow-up visit to the study site 49 days after taking their last dose for a health check-up.

This study will include participants who are healthy and will gain no benefit from taking emodepside. However, the results of the study will provide useful information to support the further development of the new emodepside tablet. The results will also provide information on the emodepside doses to be used in patients who need treatment with emodepside. Participants will be closely monitored by the study doctors for any medical problems.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 55 years of age inclusive, at the time of signing the informed consent, non-smokers, body mass index within the range of 18.0 - 29.9 kg/m2 (inclusive) at Screening
* Women that are not breastfeeding and are of non-childbearing potential aged 18 to 55 years of age inclusive, at the time of signing the informed consent, non-smokers, body mass index within the range of 18.0 - 29.9 kg/m2 (inclusive) at Screening
* Participants must be overtly healthy as determined by medical evaluation including medical history, physical examination, ECG, vital signs, and laboratory tests.
* Ability to understand and follow study-related instructions.

Exclusion Criteria:

* Medical disorder, condition or history of such that would impair the participant's ability to take part in or complete this study
* History of relevant eye or vision disorders (except myopia and hyperopia).
* History of diabetes mellitus or abnormalities in glucose homeostasis.
* Surgery, medical condition, or diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study intervention(s) will not be normal
* Febrile illness within 2 weeks before the start of the first study intervention.
* Regular use of prescription drugs, over-the-counter drugs, supplements or herbal products.
* Use of any systemic or topical medicines or substances within 2 weeks or 5 half-lives (whichever is longer) before the start of the first administration until follow-up, in particular, use of CYP3A4 inducers (including St John's Wort) or inhibitors.
* Clinically relevant findings in the physical examination and vital signs (systolic blood pressure below 90 or above 140 mmHg, diastolic blood pressure below 60 or above 90 mmHg, pulse rate below 50 or above 90 beats per minute, as measured at screening).
* Clinically relevant deviations of safety laboratory parameters in clinical chemistry, hematology, or urinalysis from reference ranges at screening.
* Suspicion of drug or alcohol abuse.
* Lack of compliance with study restrictions.
* Any vaccination received or planned during the period between 15 days before the first administration of study intervention and the last study visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) (0-72 hrs) | 0-72 hrs post dose (per period)
  • To investigate the pharmacokinetics (PK) including
  * relative bioavailability of Formulation B of emodepside (BAY 44-4400) in comparison to Formulation A
  * food-effect on Formulation B of emodepside (BAY 44-4400) If a relevant carry-over is observed in any participant as defined by C0/Cmax > 5%, corrected Cmax parameters accounting for carry-over will be calculated for all participants in addition.
Area under the concentration vs. time curve from zero to infinity after single dose (AUC) (0-72 hrs) | 0-72 hrs post dose (per period)
  • To investigate the pharmacokinetics (PK) including - relative bioavailability of Formulation B of emodepside (BAY 44-4400) in comparison to Formulation A
  - food-effect on Formulation B of emodepside (BAY 44-4400) If a relevant carry-over is observed in any participant as defined by C0/Cmax > 5%, corrected AUC parameters accounting for carry-over will be calculated for all participants in addition.

SECONDARY OUTCOMES:
Number of participants who experienced treatment-emergent adverse events (TEAEs) | After first administration of study intervention through study completion, an average of 12 weeks
  To investigate and evaluate the safety and tolerability of single oral doses of emodepside formulations in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- NUVISAN GmbH Neu-Ulm, Neu-Ulm, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the NCT number or Bayer Study ID in the search field. — https://clinicaltrials.bayer.com/study/22534